CLINICAL TRIAL: NCT04605575
Title: A Single-arm, Multi-center Phase II Clinical Study of Pyrotinib Combined With Vinorelbine in the Treatment of HER2-positive and Treated Metastatic Breast Cancer
Brief Title: Pyrotinib Plus Vinorelbine in Participants With HER2-positive Previously Treated Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wang shusen, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-002
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Pyrotinib; Breast Diseases; Vinorelbine; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — pyrotinib; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib plus vinorelbine (Experimental)
  Interventions: Drug: Pyrotinib 320mg + Vinorelbine; Drug: Pyrotinib 400mg + Vinorelbine; Drug: Pyrotinib plus Vinorelbine

INTERVENTIONS:
Drug: Pyrotinib 320mg + Vinorelbine — pyrotinib 320mg tablets administered daily by mouth, vinorelbine(po) 80 mg/m2 weekly (following a first cycle at 60 mg/m2) administered on day 1 and day 8 of 21 day cycle. Treatment lasts for two cycles
Drug: Pyrotinib 400mg + Vinorelbine — pyrotinib 400mg tablets administered daily by mouth, vinorelbine(po) 80 mg/m2 weekly (following a first cycle at 60 mg/m2) administered on day 1 and day 8 of 21 day cycle. Treatment lasts for two cycles
Drug: Pyrotinib plus Vinorelbine — pyrotinib administered daily by mouth（MTD）, vinorelbine(po) 80 mg/m2 weekly (following a first cycle at 60 mg/m2) administered on day 1 and day 8 of 21 day cycle, or vinorelbine(iv) 25 mg/m2 on day 1 and day 8 of 21 day cycle. Treatments will lasts until disease progression (as assessed by the investigator) or unmanageable toxicity.

SUMMARY:
The purpose of this study is to identify the highest tolerable dose of pyrotinib in combination with vinorelbine and to assess the safety and efficacy of the combination in Patients With HER2-Positive Locally Advanced or Metastatic Breast Cancer.

The study will be conducted in two parts. In the first part, testing will be done on up to 12 subjects to determine the highest tolerable dose of pyrotinib and vinorelbine in patients with advanced solid tumors. In the second part of the study, we will explore the safety and efficacy of Pyrotinib + vinorelbine in Patients With HER2-Positive Locally Advanced or Metastatic Breast Cancer Who Have Received Prior Trastuzumab-Based Therapy. Participants will be treated until disease progression (PD), unmanageable toxicity, or study termination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer
* HER2 status must be prospectively, centrally tested and be HER2-positive based on central laboratory assay results
* Prior treatment for breast cancer in the adjuvant, unresectable, locally advanced, or metastatic setting must include both a taxane, alone or in combination with another agent, and trastuzumab, alone or in combination with another agent. Patients who have previously used pertuzumab will be allowed.
* Documented progression (which occur during or after most recent treatment or within 6 months after completing of adjuvant therapy) of incurable, unresectable, locally advanced or metastatic breast cancer, defined by the investigator
* Measurable and/or nonmeasurable disease; participants with central nervous system-only disease are excluded
* Cardiac ejection fraction greater than or equal to (>/=) 50 percent (%) by either echocardiogram or multi-gated acquisition scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* History of treatment with pyrotinib
* Prior treatment with lapatinib or neratinib
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma
* History of receiving any anti-cancer drug/biologic or investigational treatment within 28 days prior to randomization except hormone therapy
* Recovery of treatment-related toxicity consistent with other eligibility criteria
* History of radiation therapy within 28 days of randomization
* Brain metastases that are untreated, symptomatic, or require therapy to control symptoms, as well as any history of radiation, surgery, or other therapy, including steroids, to control symptoms from brain metastases within 2 months (60 days) of randomization
* History of symptomatic congestive heart failure or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction or unstable angina
* Current severe, uncontrolled systemic disease (for example, clinically significant cardiovascular, pulmonary, or metabolic disease)
* Pregnancy or lactation
* Current known active infection with human immunodeficiency virus (HIV) or hepatitis C virus
* Presence of conditions that could affect gastrointestinal absorption: Malabsorption syndrome, resection of the small bowel or stomach, and ulcerative colitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS as Assessed by the Investigator | from enrollment to progression or death (for any reason), assessed up to 3 years
  Progression-Free Survival

SECONDARY OUTCOMES:
Objective Response Rate | Ratio of CR and PR in all subjects
  from enrollment to progression or death (for any reason), assessed up to 3 years
OS | from enrollment to progression or death (for any reason), assessed up to 3 years
  OS was defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang Jingmin, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma F, Ouyang Q, Li W, Jiang Z, Tong Z, Liu Y, Li H, Yu S, Feng J, Wang S, Hu X, Zou J, Zhu X, Xu B. Pyrotinib or Lapatinib Combined With Capecitabine in HER2-Positive Metastatic Breast Cancer With Prior Taxanes, Anthracyclines, and/or Trastuzumab: A Randomized, Phase II Study. J Clin Oncol. 2019 Oct 10;37(29):2610-2619. doi: 10.1200/JCO.19.00108. Epub 2019 Aug 20. PMID 31430226
- [Background] Li X, Yang C, Wan H, Zhang G, Feng J, Zhang L, Chen X, Zhong D, Lou L, Tao W, Zhang L. Discovery and development of pyrotinib: A novel irreversible EGFR/HER2 dual tyrosine kinase inhibitor with favorable safety profiles for the treatment of breast cancer. Eur J Pharm Sci. 2017 Dec 15;110:51-61. doi: 10.1016/j.ejps.2017.01.021. Epub 2017 Jan 21. PMID 28115222
- [Background] Ma F, Li Q, Chen S, Zhu W, Fan Y, Wang J, Luo Y, Xing P, Lan B, Li M, Yi Z, Cai R, Yuan P, Zhang P, Li Q, Xu B. Phase I Study and Biomarker Analysis of Pyrotinib, a Novel Irreversible Pan-ErbB Receptor Tyrosine Kinase Inhibitor, in Patients With Human Epidermal Growth Factor Receptor 2-Positive Metastatic Breast Cancer. J Clin Oncol. 2017 Sep 20;35(27):3105-3112. doi: 10.1200/JCO.2016.69.6179. Epub 2017 May 12. PMID 28498781